CLINICAL TRIAL: NCT04343378
Title: Prediction of Abatacept Discontinuation Using Test Reflecting Immunological Remission in Rheumatoid Arthritis
Acronym: PADIRRA
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/291/OB
Record Dates: First submitted 2020-01-09; First posted 2020-04-13 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis
Keywords: therapy discontinuation
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum; PAXgene tubes, cellular samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of this study is to identify a panel of immunological molecular and cellular biomarkers able to predict the success of major dose-reduction or discontinuation of abatacept in rheumatoid arthritis patients

DETAILED DESCRIPTION:
Parameters studied at different time points (before initiation of abatacept if sample is available in our biocollection; prior to dose tapering; prior to discontinuation) ACPA (anti-citrullinated proteins antibodies) repertoire

-IgG (Immunoglobulins G) and/or IgA auto-antibodies repertoire directed against major epitopes of well-known autoantigens

B cell repertoire B cell repertoire and transcriptome of regulatory B lymphocytes, memory B cells and B cells targeting specific autoantigens.

Analysis of type I interferon signature Expression levels of 7 type I interferon (IFN) response genes will be determined to calculate on type I IFN score

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis (RA) patients (> pr = 18 years) fulfilling the 2010 ACR/EULAR criteria
* Associated to high levels (> 3 x upper limit of normal in UA/ml) of ACPA measured by the usual anti-CCP(cyclic citrullinated proteins)2 test at the start of abatacept treatment
* Receiving IV (intravenous) or SC (subcutaneous) abatacept alone or in combination with a conventional Disease Modyfying AntiRheumatic Drugs (cDMARD) (methotrexate, leflunomide, sulfasalasin in monotherapy or in combination) according to the usual scheme or in tapering phase
* Without intra-articular injections of corticosteroids during the last 6 months prior to down-titration of abatacept
* Having discontinued corticosteroids at he time of entrance in the study
* In deep remission (Disease Activity Score (DAS) 28 ESR (or CRP) < 2.6 without clinical synovitis) since at least 1 year
* In sonographic remission at the time of enrollment (absence of PD (Power Doppler)-positive synovitis on 28 joints defined by a score < 2 on a 0-3 semi-quantitative scale for each joint)

Exclusion Criteria:

* Age < 18 years
* RA negative for ACPA (anti-citrullinated proteins antibodies) or not fulfilling ACR/EULAR criteria
* Abatacept discontinuation due to serious adverse event, loss of efficacy or pregnancy project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ACPA + RA patients from the rheumatology department of Rouen University Hospital receiving IV (intravenous) or SC (subcutaneous) abatacept (according to the usual scheme or having started tapering) and in deep remission (as defined previously) will be included.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
relapse | from date of inclusion until the date of documented flare assessed up to 24 months
  Increase of DAS(Disease Activity Score)28 ESR (or CRP) > 3.2 at 2 consecutive time points.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier VITTECOQ, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No